CLINICAL TRIAL: NCT01924650
Title: A Randomized, Open Label, Single Dose, 6 Treatment, 4-way Crossover Study in Healthy Subjects to Assess the Pharmacokinetics of Three Different Particle Sizes of PH-797804 Tablet With and Without the Solubilizing Agent Sodium Lauryl Sulphate (SLS)
Brief Title: A Pharmacokinetic Study of Three Different Particle Sizes of PH-797804
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6631040
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
MeSH Terms: interventions — PH 797804

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- PH-797804 PARTICLE SIZE 9-11UM (Experimental)
  Interventions: Drug: PH-797804
- PH-797804 PARTICLE SIZE 9-11UM WITH SLS (Experimental)
  Interventions: Drug: PH-797804
- PH-797804 PARTICLE SIZE <= 20UM (Experimental)
  Interventions: Drug: PH-797804
- PH-797804 PARTICLE SIZE <= 20UM WITH SLS (Experimental)
  Interventions: Drug: PH-797804
- PH-797804 PARTICLE SIZE <= 5UM (Experimental)
  Interventions: Drug: PH-797804
- PH-797804 PARTICLE SIZE <= 5UM WITH SLS (Experimental)
  Interventions: Drug: PH-797804

INTERVENTIONS:
Drug: PH-797804 — Tablet, 6 mg, single dose
  Arms: PH-797804 PARTICLE SIZE 9-11UM
Drug: PH-797804 — Tablet, 6 mg, single dose
  Arms: PH-797804 PARTICLE SIZE 9-11UM WITH SLS
Drug: PH-797804 — Tablet, 6 mg, single dose
  Arms: PH-797804 PARTICLE SIZE <= 20UM
Drug: PH-797804 — Tablet, 6 mg, single dose
  Arms: PH-797804 PARTICLE SIZE <= 20UM WITH SLS
Drug: PH-797804 — Tablet, 6 mg, single dose
  Arms: PH-797804 PARTICLE SIZE <= 5UM
Drug: PH-797804 — Tablet, 6 mg, single dose
  Arms: PH-797804 PARTICLE SIZE <= 5UM WITH SLS

SUMMARY:
The purpose of this study is to investigate the effects of varying particle size on the pharmacokinetics of PH-797804

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and/or healthy female subjects of non-child bearing potential between the ages of 18 and 55 years (inclusive). Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurements, 12-lead ECG and clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight > 50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 drinks/week for males.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Time 72 hours (AUC72) | 0,2,3,4,5,6,8,12,24,48,72 hours post-dose
  Area under the plasma concentration time-curve from zero to 72 hours (AUC72)
Maximum Observed Plasma Concentration (Cmax) | 0,2,3,4,5,6,8,12,24,48,72 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 0,2,3,4,5,6,8,12,24,48,72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6631040&StudyName=A%20Pharmacokinetic%20Study%20of%20Three%20Different%20Particle%20Sizes%20of%20PH-797804